CLINICAL TRIAL: NCT07229911
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Sponsor-Open Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-781 in Healthy Participants and a Single-Arm, Open-Label Evaluation in Participants With Non-Cirrhotic Primary Sclerosing Cholangitis
Brief Title: A Study of TAK-781 in Healthy Volunteers and in Participants With Non-Cirrhotic Primary Sclerosing Cholangitis (PSC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-781-1001
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Primary Sclerosing Cholangitis
Keywords: Drug Therapy
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 1a will be double blind, whereas Phase 1b will be non-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Phase 1a (Part 1): TAK-781 SAD (Experimental): Healthy participants will receive a single dose of TAK-781 injection at different dose level cohorts (1-6) on Day 1 of the pre-defined treatment period. An additional cohort may be added to repeat a selected dose from one of the previously tested dose levels in order to assess safety and tolerability and/or to verify the level of target engagement (TE).
  Interventions: Drug: TAK-781
- Phase 1a (Part 1): Placebo SAD (Placebo Comparator): Healthy participants will receive TAK-781 matching placebo injection on Day 1 of the pre-defined treatment period.
  Interventions: Drug: Placebo
- Phase 1a (Part 2): TAK-781 MAD (Experimental): Healthy participants will receive multiple doses of TAK-781 injection across five cohorts (1 to 5), with or without a loading dose during the pre-defined treatment period. An additional cohort may be added to repeat a selected dose level and/or dosing regimen from one of the previously tested dose levels and/or dosing regimens in order to assess safety and tolerability, and/or to verify the level of TE.
  Interventions: Drug: TAK-781
- Phase 1a (Part 2): Placebo MAD (Placebo Comparator): Healthy participants will receive multiple doses of TAK-781 matching placebo injection, with or without a loading dose during the pre-defined treatment period.
  Interventions: Drug: Placebo
- Phase 1b (Part 3): TAK-781 (Experimental): Participants with non-cirrhotic PSC will receive a single dose of TAK-781 injection on Day 1 during the pre-defined treatment period. Part 3 will not begin until the SAD portion of the trial is considered complete.
  Interventions: Drug: TAK-781

INTERVENTIONS:
Drug: TAK-781 — TAK-781 injection.
  Arms: Phase 1a (Part 1): TAK-781 SAD; Phase 1a (Part 2): TAK-781 MAD; Phase 1b (Part 3): TAK-781
Drug: Placebo — TAK-781 matching placebo injection.
  Arms: Phase 1a (Part 1): Placebo SAD; Phase 1a (Part 2): Placebo MAD

SUMMARY:
The main aim of this study is to see if the drug TAK-781 is safe for healthy volunteers and for participants with PSC. The study will also look at how well participants can tolerate TAK-781. In addition, the study will check how the body absorbs, uses, and gets rid of TAK-781 (Pharmacokinetics [PK]), how the drug affects the body (Pharmacodynamics [PD]), and how the body's immune system reacts to TAK-781 (Immunogenicity).

The study consists of two phases (Phase 1a and 1b). Phase 1a includes two parts: Part 1 (Single Ascending Dose [SAD]) and Part 2 (Multiple Ascending Dose [MAD]). In Part 1, healthy participants will receive either single dose of TAK-781 or a placebo. A placebo looks the same as TAK-781 but has no medicine in it. In Part 2, healthy participants will receive multiple doses of TAK-781 or a placebo. In Phase 1b (Part 3), participants with large duct, non-cirrhotic PSC will receive a single dose of TAK-781.

Participants will be in the study for about 36 weeks.

ELIGIBILITY:
Inclusion Criteria: Phase 1a (SAD and MAD)

1. The participant is willing and able to fully comply with all trial procedures and requirements, in the investigator's opinion.
2. The participant has provided informed consent (that is, in writing, documented via a signed and dated informed consent form (ICF) or electronic consent [e-consent] if applicable) and any required privacy authorization prior to the initiation of any trial procedures.
3. Male at birth and female at birth participants aged 18 to 68 years, inclusive, at the time of consent.
4. The participant is judged to be in good health (for example, no evidence of cardiovascular, liver, metabolic, gastroenterological, or kidney disease) by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, ECG, and vital sign measurements performed at the first screening visit.
5. The participant must have a body mass index (BMI) of less than 30.0 kilograms per square meter (kg/m^2) at the time of screening.
6. Has not had frequent or heavy use (that is, near-daily) of medical or recreational cannabis for at least 3 months before screening.
7. The participant must not be a person of childbearing potential (POCBP) defined by at least 1 of the following criteria:

   * Surgically sterile for at least 6 weeks at screening (defined as having undergone one of the following procedures: hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).
   * Postmenopausal at screening (defined as no menses for 12 months without an alternative medical cause). A high follicle-stimulating hormone (FSH) level (greater than or equal to [>=]40 international units/liter [IU/L] in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
   * Has no uterus as a result of congenital condition. The participant must not donate ova for at least 6 months after the last dose of trial intervention.
8. Male participants (based on sex at birth) must use highly effective contraception, from the date of signing the ICF, throughout the duration of the trial, and for 6 months after the last dose of trial intervention. The participant must not donate sperm for at least 6 months after the last dose of trial intervention.

Inclusion Criteria: Phase 1b (Non-Cirrhotic PSC)

1. The participant is willing and able to fully comply with all trial procedures and requirements, in the investigator's opinion.
2. The participant has provided informed consent (that is, in writing, documented via a signed and dated ICF or e-consent if applicable) and any required privacy authorization prior to the initiation of any trial procedures.
3. Male at birth and female at birth participants aged 18 to 68 years, inclusive, at the time of consent.
4. Confirmed diagnosis of large-duct PSC based on any 2 of the following 3 criteria:

   * Historical evidence of an elevated alkaline phosphatase (ALP) greater than [>] upper limit of normal (ULN) from any laboratory.
   * Historical liver biopsy with histologic features consistent with large-duct PSC, in the appropriate clinical context (such as cholestatic liver enzyme profile, inflammatory bowel disease [IBD] history).
   * Historical abnormal cholangiography consistent with PSC as measured by magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography, or percutaneous transhepatic cholangiography.
5. The participants must have a fibrogenesis biomarker over pre-defined level.
6. The participants must have evidence for moderate/advanced fibrosis but not cirrhosis as defined by enhanced liver fibrosis (ELF) >= 7.7 but less than or equal to (<=) 11.3 at Visit 1.
7. No evidence of cholangiocarcinoma or any other malignancy on magnetic resonance imaging (MRI) at screening.
8. Participants with a certain concomitant disease are allowed to enroll if pre-defined criteria are met.
9. Participants must have certain additional laboratory parameters in specified ranges at screening.
10. Has not had frequent or heavy use (that is, near-daily) of medical or recreational cannabis for at least 3 months before screening.
11. A female and male participant (based on sex at birth) must use highly effective contraception, from the date of signing the ICF, throughout the duration of the trial, and for 6 months after the last dose of trial intervention. The participant must not donate ova or sperm for at least 6 months after the last dose of trial intervention.
12. A POCBP must have a negative serum pregnancy test at first screening visit and urine pregnancy test on second screening visit and Day 1 before dosing.
13. Participants must be able to be educated regarding the correct process/procedure, verbally state understanding and comply with the correct process/procedure of the administration SC investigational product (IP) for the duration of the trial.

Exclusion Criteria: Phase 1a (SAD and MAD)

1. The participant is an employee of the sponsor or trial site, or an immediate family member (for example, spouse, parent, child, sibling) of an employee of the sponsor or trial site who is directly involved in the conduct of the trial.
2. The participant has a known hypersensitivity to any component of the formulation of TAK-781 or related compounds.
3. The participant has a history of significant multiple and/or severe allergies (for example, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
4. The participant has a history or clinical evidence of bleeding diathesis or any coagulation disorder.
5. The participant has a medical history of prior cholecystectomy.
6. The participant has participated in another investigational trial with other investigational agents or devices for any indication within 4 weeks or within 5 half-lives, for investigational drugs or biologics with a known half-life (whichever is longer), before the screening visit. The interval window from the previous trial will be derived from the date of the last trial medical procedure, and/or AE related to the trial IP or procedure in the previous trial to the screening visit of the current trial. Exceptions may be made for observational, natural history and nonintervention type studies with sponsor or designee approval.
7. The participant has an ALT and/or AST value greater than the ULN during screening.
8. The participant has abnormal cholesterol: total cholesterol >200 milligrams per deciliter (mg/dL), low-density lipoprotein cholesterol (LDL-c) (>100 mg/dL), high-density lipoprotein cholesterol (HDL-C) (lesser than [<]45 mg/dL for male, <55 mg/dL for female), and triglycerides (>150 mg/dL) at screening.
9. The participant has eGFR rate <= 90milliliter per minutes per 1.73 square meters (mL/min/1.73m^2) at screening.
10. The participant screening ECG (triplicate) reveals a QT interval with Fridericia correction method (QTcF) > 450 millisecond (ms) (male) or > 460 ms (female).
11. The participant has a history of torsades de pointes, ventricular rhythm disturbances (for example, ventricular tachycardia), heart block (excluding first-degree block, being PR interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on ECG.
12. The participant has a confirmed supine systolic blood pressure >= 130 millimetres of mercury (mmHg) and/or diastolic blood pressure >=90 mmHg at screening. If the participant's supine blood pressure exceeds these thresholds, the measurement should be repeated twice after the participant has remained in the supine position for at least 10 minutes. The average of the three supine blood pressure measurements will be used to determine eligibility.

    Resting BP is defined as a BP measurement obtained after the participant has been resting for a minimum of 5 minutes.
13. The participant has a resting heart rate (HR) outside of the range of 55 to 100 beats per minute (bpm) (inclusive) at screening, confirmed on repeat testing within a maximum of 30 minutes. Athletic participants with HR <55 bpm may be enrolled based on the investigator's judgement provided that the HR is >45 bpm.
14. The participant has a positive urine screen for drugs of abuse at screening and Day -3.
15. History of any malignancy diagnosed or treated within 5 years prior to screening.
16. The participant consumes excessive amounts (defined as greater than 600 milligram (mg) of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
17. Has a positive pregnancy test result during the screening period.
18. Participants who test negative for hepatitis B surface antigen (HBsAg) but positive for hepatitis B core antibody (HBcAb) would be considered eligible if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) results are negative at screening (as confirmed by HBV DNA polymerase chain reaction [PCR] reflex testing performed by the central laboratory). Participants with positive HBV DNA test results will not be eligible.
19. Participants who test positive for hepatitis C virus (HCV) ribonucleic acid (RNA) at screening. Participants who are hepatitis C antibody (HCVAb) positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks before screening Visit 1]).
20. The participant tests positive for human immunodeficiency virus (HIV) at screening or currently receiving antiretroviral therapy.
21. Has undergone major surgery or donated or lost 1 unit of blood (approximately 500 milliliters [mL]) within 4 weeks before the screening visit.
22. Currently has or previously had a significant illness, as judged by the investigator, within 2 weeks of the first dose of trial intervention.
23. The participant is unable to refrain from or anticipates using prohibited or excluded medications, herbal preparations, grapefruit juice, and other restricted substances or the required washout period prior to administration of the first dose of trial intervention throughout the trial and until the follow-up visit.
24. The participant is unable to refrain from or anticipate using smoking, vaping or nicotine-containing products 2 weeks before screening until the last follow-up visit.
25. Clinically relevant drug or alcohol abuse within 12 months of screening.

    * A positive drug screen is exclusive unless it can be explained by a prescribed medication.
    * Participant with alcohol consumption greater than 4 units on any day or 14 units per week for male participants, or greater than 3 units on any day or 7 units per week for female participants [1 unit of alcohol is present in one 12 ounce (oz)/355 mL beer (approximately 5 percent (%) alcohol), one 5 oz/148 mL glass of wine (approximately 12% alcohol), and one 1.5 oz/44 mL measure of 80-proof liquor (approximately 40% alcohol)].

Exclusion Criteria: Phase 1b (Non-Cirrhotic PSC)

1. Presence of documented secondary sclerosing cholangitis (such as ischemic cholangitis, recurrent pancreatitis, intraductal stone disease, severe bacterial cholangitis, surgical or blunt abdominal trauma, recurrent pyogenic cholangitis, cholelithiasis, choledocholithiasis, toxic sclerosing cholangitis due to chemical agents, or any other cause of secondary sclerosing cholangitis) on prior clinical investigations.
2. Immunoglobulin G4-related Sclerosing Cholangitis based on historical diagnosis.
3. Evidence of compensated cirrhosis. All participants will undergo a standardized cirrhosis exclusion assessment during screening including clinical, laboratory, and imaging evaluation (non-contrast MRI/ magnetic resonance elastography [MRE], MRCP+), documented using a predefined cirrhosis checklist completed and signed by both the site Principal Investigator (or Sub-Investigator) and the site radiologist. For participants with ELF >9.8 to <= 11.3 and/or liver stiffness measurement (LSM) >12.5 kilopascals (kPa), the checklist findings will undergo enhanced review by the sponsor medical monitor, who will provide final eligibility confirmation. A hepatic adjudication committee may be consulted in cases of ambiguity or disagreement. Participants will be excluded if >= 2 of the following cirrhosis-associated features are present:

   * MRE liver stiffness >= 4.32 kPa.
   * Liver surface nodularity or lobar redistribution.
   * Spleen volume >400 mL/m^2 body surface area or spleen length >13 centimeter (cm).
   * Segmental parenchymal signal heterogeneity, periportal edema, or lobar atrophy.
   * Collateral vessels or signs of portal hypertension (for example, varices, recanalized umbilical vein).
   * Radiologist overall impression consistent with cirrhosis.
   * Serum albumin <3.5 grams per deciliter (g/dL).
4. The participant has a medical history of prior cholecystectomy.
5. Participants will be excluded if they meet any of the following criteria: a diagnosis of decompensated liver disease, or evidence of new signs of decompensation or clinically meaningful deterioration in liver function during the screening period, based on the judgment of the investigator. This may include, but is not limited to, significant changes in the following parameters: total bilirubin, direct bilirubin, albumin, international normalized ratio (INR), creatinine, alanine transaminase (ALT), or aspartate transaminase (AST).
6. Presence or history of any of the following:

   * Ascites.
   * Hepatic encephalopathy.
   * Variceal bleeding.
   * Child-Pugh score >6 (Class B or C), unless elevated INR is attributable to therapeutic anticoagulation. (Participants with compensated cirrhosis [for example, Child-Pugh A] will also be excluded if identified via the noninvasive cirrhosis exclusion algorithm, which includes assessment of ELF score, LSM, MRI/MRE, MRCP+, and clinical/laboratory parameters).
   * Model for End-Stage Liver Disease score >11.
7. Concomitant overlap syndrome with autoimmune hepatitis as diagnosed at screening by AST or ALT > 5 * ULN, and historical:

   * Positive smooth muscle antibody and/or liver-kidney microsomal antibody (LKM), or
   * Immunoglobulin G (IgG) >ULN, or
   * Biopsy suggestive for autoimmune hepatitis.
8. Concomitant overlap syndrome with primary biliary cholangitis (PBC) as diagnosed by either historical:

   * Positive anti-mitochondrial autoantibodies, or
   * Biopsy suggestive for PBC.
9. Clinically significant acute or chronic liver disease of an etiology other than PSC.
10. Presence of a dominant stricture of clinical concern on MRCP at screening. However:

    - Participants with dominant stricture could be enrolled if the investigator determines that there is no evidence on MRI or cholangiography indicative of cholangiocarcinoma or that the stricture will likely not result in significant fluctuations in ALP during screening or trial period.
11. Placement of a bile duct stent or percutaneous bile duct drain within 3 months of screening. However:

    - Participants who had undergone a stricture balloon dilation procedure can enroll in the trial after at least 4 weeks post procedure.
12. History, evidence, or high suspicion of cholangiocarcinoma or other hepatobiliary malignancy based on imaging, laboratory values, and/or clinical symptoms.
13. Ascending cholangitis within 60 days prior to screening and through Day 1. However:

    * Chronic preventive antibiotics for cholangitis are allowed in the trial.
    * Intermittent courses of antibiotics for the presumptive treatment of cholangitis are allowed if outside the 12-week window prior to screening.
14. Prior liver transplantation.
15. Screening ECG with clinically significant abnormalities as determined by the investigator.
16. Participants who test negative for HBsAg but positive for HBcAb would be considered eligible if HBV DNA results are negative at screening (as confirmed by HBV DNA PCR reflex testing performed by the central laboratory). Participants with positive HBV DNA test results will not be eligible.
17. Participants who test positive for HCV RNA at screening. Participants who are HCVAb positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks before baseline]).
18. The participant tests positive for HIV at screening or currently receiving antiretroviral therapy.
19. History of malignancy diagnosed or treated within 5 years prior to screening.
20. The participant is unable to refrain from or anticipates using prohibited or excluded medications, herbal preparations, grapefruit juice, and other restricted substances or the required washout period prior to administration of the first dose of trial intervention throughout the trial and until the follow-up visit.
21. The participant has not had frequent or heavy use (>= 20 cigarettes per day) of smoking, vaping or nicotine-containing products or has not smoking-related complications.
22. Clinically relevant drug or alcohol abuse within 12 months of screening.

    * A positive drug screen is exclusive unless it can be explained by a prescribed medication.
    * Participant with alcohol consumption greater than 4 units on any day or 14 units per week for male participants, or greater than 3 units on any day or 7 units per week for female participants [1 unit of alcohol is present in one 12 oz/355 mL beer (approximately 5% alcohol), one 5 oz/148 mL glass of wine (approximately 12% alcohol), and one 1.5 oz/44 mL measure of 80-proof liquor (approximately 40% alcohol)].
23. Use of any prohibited concomitant medication is not allowed unless the participant has completed the washout period prior to Day 1.
24. Participants should not be currently taking ursodeoxycholic acid, unless they have completed the washout period prior to Day 1.
25. Severe allergic or anaphylactic reactions to any components of N-acetylgalactosamine small-interfering RNA therapeutics.
26. Use of any investigational drug, biologic, or medical device, or participation in an interventional clinical trial, is prohibited within 4 weeks prior to screening or within 5 elimination half-lives for investigational drugs or biologics with a known half-life (whichever is longer). This restriction includes any pharmacologic, endoscopic, or other interventional procedures intended to modify or alter the course of PSC or its underlying disease processes.
27. History of clinically significant unstable or untreated illness or any other major medical disorder that may have interfered with participant treatment, assessment, or compliance with the protocol.
28. Any acute or chronic condition or other disease that, in the opinion of the investigator, would limit the ability of the participant to complete and/or participate in the clinical trial.
29. Presence of any other conditions (for example, geographic or social), actual or projected, that the investigator determines would restrict or limit the participation of the participant for the duration of the trial.
30. Individuals who are employed by the sponsor, a participating contract research organization (CRO), or the trial site - including permanent staff, temporary or contract workers, or designees directly involved in the conduct of the trial - are excluded from participation. This exclusion also applies to immediate family members (defined as spouse, parent, child, or sibling, whether biological, adoptive, or legally recognized) of employees of the sponsor, CRO, or trial site. For large university or academic health systems, this restriction applies only to individuals who are directly involved in the conduct or oversight of the clinical trial or who are part of the same department/unit conducting the trial, in order to minimize conflict of interest.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2028-04-06 (Estimated); Study Completion 2028-04-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1a (SAD and MAD) and Phase 1b: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Phase 1a (SAD) and 1b: From start of study drug administration up to End of Treatment (EOT)/Early termination (ET) (up to Week 20); Phase 1a (MAD): From start of study drug administration up to EOT/ET (up to Week 32)
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a trial intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the trial intervention.
Phase 1a (SAD and MAD) and Phase 1b: Number of Participants With Clinically Significant Changes in Clinical Laboratory Values | Phase 1a (SAD) and 1b: From start of study drug administration up to EOT/ET (up to Week 20); Phase 1a (MAD): From start of study drug administration up to EOT/ET (up to Week 32)
  Laboratory parameters will include hematology, chemistry and urinalysis. Any clinically significant change in laboratory values will be determined at the investigator's discretion.
Phase 1a (SAD and MAD) and Phase 1b: Number of Participants With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) Parameters | Phase 1a (SAD) and 1b: From start of study drug administration up to EOT/ET (up to Week 20); Phase 1a (MAD): From start of study drug administration up to EOT/ET (up to Week 32)
  The 12-lead ECG will be evaluated. Any clinically significant change in ECG assessment will be determined at the investigator's discretion.
Phase 1a (SAD and MAD) and Phase 1b: Number of Participants With Clinically Significant Changes in Vital Sign Values | Phase 1a (SAD) and 1b: From start of study drug administration up to EOT/ET (up to Week 20); Phase 1a (MAD): From start of study drug administration up to EOT/ET (up to Week 32)
  Vital signs will include measurement of oral body temperature, supine blood pressure and heart rate. Any clinically significant change in vital signs will be determined at the investigator's discretion.

SECONDARY OUTCOMES:
Phase 1a and 1b: Maximum Observed Plasma Concentration (Cmax) of TAK-781 | Predose up to 2 days post-dose
  Cmax of TAK-781 will be reported.
Phase 1a and 1b: Time of First Occurrence of Plasma Cmax (Tmax) of TAK-781 | Predose up to 2 days post-dose
  Tmax of TAK-781 will be reported.
Phase 1a and 1b: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUCinf) of TAK-781 | Predose up to 2 days post-dose
  AUCinf of TAK-781 will be reported.
Phase 1a and 1b: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUClast) of TAK-781 | Predose up to 2 days post-dose
  AUClast of TAK-781 will be reported.
Phase 1a: Percentage Change From Baseline in TE Biomarker Area Under the Effect Curve 0 to 9 Hours (AUEC0-9h) | Phase 1a: 0 to 9 hours post-dose
  Percentage change from baseline in TE biomarker AUEC0-9h will be reported.
Phase 1b: Percentage Change From Baseline in Fibrogenesis Biomarker Levels | Baseline up to Week 12
  Percentage change from baseline in fibrogenesis biomarker levels will be reported.
Phase 1b: Percentage Change From Baseline in TE Biomarker Through Week 12 | Baseline up to Week 12
  Percentage change from baseline in TE biomarker through Week 12 will be reported.
Phase 1a (SAD and MAD) and 1b: Number of Participants With Anti-drug Antibodies (ADAs) to TAK-781 | Phase 1a (SAD) and 1b: Baseline up to Week 20; Phase 1a (MAD): Baseline up to Week 32
  Number of participants with ADAs to TAK-781 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- ICON, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/ecc353299a5c4a7b??page=1&idFilter=TAK-781-1001